CLINICAL TRIAL: NCT06146647
Title: Dove Self-Esteem Project: Evaluating Effectiveness and Acceptability of Two Positive Body Image Micro-interventions on Young Children's Body Functionality Appreciation, State Body Appreciation and Anti-fat Attitudes
Brief Title: The Evaluation of Two Positive Body Image Micro-interventions for Children Aged 4-6 Years
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DSEP_GOOSE
Record Dates: First submitted 2023-11-15; First posted 2023-11-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Body Image; Anti Fat Bias
Keywords: weight stigma; anti-fat bias; body appreciation; body functionality; body satisfaction; body dissatisfaction; children's media; music video; body image
MeSH Terms: conditions — Weight Prejudice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Masking is not possible for the investigator due to the trial design and protocol for data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention condition: 15 minute (approx.) show with positive body image messaging (Experimental): Those assigned to this arm will watch the 15 minute tv show with positive body image content.
  Interventions: Behavioral: Positive body image TV show
- Control condition: 15 minute (approx.) show without positive body image messaging (Active Comparator): Those assigned to this condition will watch a 15 minute tv show that does not contain positive body image content.
  The show that will be used for this condition is about a tv character visiting the dentist.
  Interventions: Behavioral: Active control TV show about a visit to the dentist
- Intervention condition: Music video with positive body image messaging (Experimental): Those assigned to this condition will watch the music video containing positive body image messaging.
  Interventions: Behavioral: Positive body image music video
- Control condition: Music video without positive body image content (Active Comparator): Those assigned to this condition will watch a music video without positive body image messaging.
  The music video that will be used for this condition is about brushing teeth.
  Interventions: Behavioral: Active control music video about brushing teeth

INTERVENTIONS:
Behavioral: Positive body image TV show — This is a 15 minute (approximately) show that has positive body image content embedded in the storyline. It also showcases a diverse range of body sizes in the casting.
  Arms: Intervention condition: 15 minute (approx.) show with positive body image messaging
Behavioral: Positive body image music video — This is a positive body image song with strong visual representation of diverse body sizes in the music video.
  Arms: Intervention condition: Music video with positive body image messaging
Behavioral: Active control TV show about a visit to the dentist — 14 minute tv show following a tv character as he visits the dentist.
  Arms: Control condition: 15 minute (approx.) show without positive body image messaging
Behavioral: Active control music video about brushing teeth — Music video of a tv character singing about brushing teeth
  Arms: Control condition: Music video without positive body image content

SUMMARY:
The goal of this 4-arm randomized controlled trial is to test the effectiveness of two positive body image media micro interventions (a tv show and a music video) in improving body image related constructs.

The main questions this study aims to answer are:

1. Relative to time-matched active controls, are the two positive body image media micro-interventions effective in yielding immediate improvements in children's body functionality appreciation and body appreciation and in reducing anti-fat attitudes?
2. Are the two positive body image media micro-interventions acceptable to children and their participating parent/guardian?

An additional five secondary exploratory research questions are described below [in the description section].

Participants will be recruited into the trial by a research agency via their parents/guardians. Once recruited, they will be randomised into one of 4 conditions:

* 15-minute TV intervention
* 15-minute active TV control
* 3-minute music video intervention
* 3-minute active music video control

Children (and their parent or guardian) will visit a testing centre in groups of approximately 12 dyads. Children will complete T1 assessment interviews one-on-one with a researcher, before watching their assigned media with their parent. After watching their assigned media, children will complete their T2 assessment, again one-to-one with a researcher, while parents complete a survey regarding their acceptability of the media they watched. Parents/guardians will be given a link to rewatch their assigned media and encouraged to rewatch with their child before returning to the testing centre approximately one week later. When children and parents/guardians return one week later, the child will complete T3 assessment interviews one-to-one with a researcher, and parents will complete a short survey regarding their rewatch habits.

Researchers will compare the two positive body image media micro-interventions with their time-matched active controls to examine if they are effective in yielding immediate improvements in children's body functionality appreciation and body appreciation and in reducing anti-fat attitudes.

DETAILED DESCRIPTION:
Body Image in Childhood

Body image develops in early childhood (Grogan et al., 2021) and by age four children report negative feelings towards their body and negative attitudes (e.g., anti-fat bias) towards others (Bensley et al., 2023; Paxton & Damiano, 2017). Body image concerns are associated with low self-esteem, disordered eating and academic disengagement (Bornioli et al., 2019) as children emerge into adolescence. As such, it is important to intervene and implement age-appropriate prevention strategies as early as possible. One key prevention strategy, endorsed by scholars and body image experts (e.g., Daniels & Roberts, 2018), is to foster positive body image among children through the development and evaluation of interventions.

Children's Media

Children's media has proven a powerful tool in educating young children, with countless shows designed to assist language development, moral understanding and pro-social behaviour (e.g., Sesame Street; Fisch & Truglio (2014), Daniel's Tiger; Rasmussen et al., 2016). However, only a small portion of these have undergone rigorous scientific evaluation and even fewer target positive body image. One study evaluated short-animated stories targeting risk and protective factors for body image among 7 - 10 year olds and found improvements in state body satisfaction, trait media literacy and pro-social behaviours with effects maintained at 1-week follow-up (Matheson et al., 2020). Other successful media-based approaches among older demographics have included online games (e.g., Matheson et al, 2022), e-books (e.g., Matheson et al., in prep) and traditional board games (e.g., Guest et al., 2021).

The Current Interventions

The positive body image media micro-interventions to be evaluated are currently being developed. The first intervention, a TV episode, centres around a talent show and teaches children to discover and love the wonderful and exciting things their bodies can do. Specifically, the episode follows the story of a young boy who wants to take part in a talent show but lacks confidence in a particular dance move. He, and some of the other talented dancers in the tv show, live in a larger body, thus disrupting traditionally held size stereotypes. The second positive body image media micro-intervention, a music video, also showcases diverse body sizes. The lyrics in the song, sung to the tune of 'Head, Shoulders, Knees and Toes', details all the amazing things our bodies can do and models the characters expressing love for their body. The content is based on existing empirical evidence, knowledge about body image and includes two main themes:

1. Body Functionality Appreciation (focusing on what the body can do rather than what it looks like).
2. Acceptance of Appearance Diversity (celebrating that everybody is different, and people come in all shapes and sizes).

This project will include a pilot study, followed by a fully powered randomised controlled trial (RCT). The purpose of the pilot study is to check the research design and protocols are fit for purpose.

Specifically, a stop/go protocol will be followed.

The research team will PROCEED to the main trial provided:

1. at least 80% of the data is considered 'usable' (based on participant attendance, non-completion, participant engagement and comprehension)
2. There is no evidence of ceiling effects for the measures at T1.
3. There is no evidence of harm (ie., child distress due to the content of the micro-interventions or the research process).

The research team will REVIEW research processes if:

1. Between 60-80% of the data is usable
2. There is some evidence of ceiling effects at T1
3. There is some evidence of participant distress (between 1-10% of participants)

The research team will NOT proceed to the main trial if:

1. Less than 60% of the data is usable
2. Every measure demonstrates ceiling effects
3. There is evidence that more than 10% of participants experience distress

Should the study proceed to a main trial, the aims, research questions and hypotheses of the main trial are as follows;

RQ1. Relative to time-matched active controls, are the two positive body image media micro-interventions effective in yielding immediate improvements in children's body functionality appreciation and body appreciation and in reducing anti-fat attitudes?

H1: The researchers anticipate children randomised into one of the interventions conditions to experience an immediate improvement (T2) in body functionality appreciation and body appreciation, relative to the control groups. The researchers also expect the intervention groups to report an immediate reduction in anti-fat attitudes (T2), relative to the control groups.

RQ2. Are the two positive body image media micro-interventions acceptable to children and their participating parent/guardian?

H2. The researchers expect the two positive body image media micro-interventions to be enjoyed by children and viewed as age appropriate and relevant by their participating parent/guardian.

Further, there are five exploratory research questions, examining moderators, exposure effects, and sustained effects:

RQ3. Does gender moderate intervention effectiveness?

H3. The researchers predict that the intervention will be more effective for girls than for boys.

RQ4. Does year group moderate intervention effectiveness?

H4. The researchers predict that the intervention will be more effective for children in year 1 than children in reception.

RQ5. Are there within-group intervention effects whereby repeated exposure to either one of the positive body image media micro-interventions is positively correlated to improvements at T3?

H5. The researchers expect that children within each intervention condition (e.g., TV and music video) will experience greater improvements to body functionality appreciation and body appreciation and greater reductions in anti-fat attitudes, at one-week follow up (T3) the more they have watched their content from T2 to T3.

RQ6. Is there a difference in terms of the immediate pre-post effectiveness outcomes between the two interventions?

H6. The researchers anticipate the 15-minute intervention will be more effective than the 2/3-minute music video on the premise that there will be greater exposure to core messaging.

RQ7. Are there sustained effects approximately one week following media exposure, controlling for repeat watching?

H7: The researchers anticipate to see sustained effects in our outcome measures at one week follow-up, relative to the control condition, controlling for repeat watching.

ELIGIBILITY:
Inclusion Criteria:

1. Child is aged 4, 5, or 6 years old
2. Child is currently in reception or Year 1 of primary school
3. The child's parent/guardian resides in Greater London or the Midlands.

Exclusion Criteria:

1. Child has complex special educational needs
2. Child is a sibling of a child already recruited into the study
3. Child is not English speaking
4. Child is home-schooled

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 440 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in body appreciation | Baseline; post-intervention (immediate post); follow-up (10 days later)
  Participants respond to two 4-point Likert scale questions, 'Do you love your body?' and 'Do you think your body is amazing?' (No, a little, bit, a medium bit, a lot)

SECONDARY OUTCOMES:
Change in anti-fat attitudes | Baseline; post intervention (immediate post); follow-up (10 days later)
  Children rate a smaller child character and a larger child character on five dimensions (e.g. is this child cute, ugly, or somewhere in the middle?). Child character to be matched as closely as possible on gender and ethnicity to participant.
Change in body functionality appreciation | Baseline; post intervention (immediate post); follow-up (approx. 10 days later)
  Participants have a minimum of 60 seconds to tell the moderator all the amazing things that they can do with their body. A frequency score will be calculated (i.e., the number of things a participant thinks there body can do that is amazing). Change will be measured as a frequency. This is a bespoke, purpose built measure.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Craddock, PhD, Principal Investigator — University of the West of England
Locations (1):
- Centre for Appearance Research, UWE, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bensley J, Riley HO, Bauer KW, Miller AL. Weight bias among children and parents during very early childhood: A scoping review of the literature. Appetite. 2023 Apr 1;183:106461. doi: 10.1016/j.appet.2023.106461. Epub 2023 Jan 13. PMID 36642116
- [Background] Guest E, Jarman H, Sharratt N, Williamson H, White P, Harcourt D, Slater A; VTCT Foundation Research Team at the Centre for Appearance Research. 'Everybody's Different: The Appearance Game'. A randomised controlled trial evaluating an appearance-related board game intervention with children aged 9-11 years. Body Image. 2021 Mar;36:34-44. doi: 10.1016/j.bodyim.2020.09.010. Epub 2020 Nov 5. PMID 33160256
- [Background] Matheson EL, Lewis-Smith H, Diedrichs PC. The effectiveness of brief animated films as a scalable micro-intervention to improve children's body image: A randomised controlled trial. Body Image. 2020 Dec;35:142-153. doi: 10.1016/j.bodyim.2020.08.015. Epub 2020 Oct 10. PMID 33049455
- [Background] Matheson, E. L., Smith, H. G., Lewis-Smith, H., Arbon, R. E., & Diedrichs, P. C. (2022). Game on! A randomised controlled trial evaluation of playable technology in improving body satisfaction and negative affect among adolescents. new media & society, 24(12), 2635-2658.
- [Background] Paxton SJ, Damiano SR. The Development of Body Image and Weight Bias in Childhood. Adv Child Dev Behav. 2017;52:269-298. doi: 10.1016/bs.acdb.2016.10.006. Epub 2016 Dec 9. PMID 28215287
- [Background] Rasmussen, E. E., Shafer, A., Colwell, M. J., White, S., Punyanunt-Carter, N., Densley, R. L., & Wright, H. (2016). Relation between active mediation, exposure to Daniel Tiger's Neighborhood, and US preschoolers' social and emotional development. Journal of Children and Media, 10(4), 443-461.
- [Derived] Smith HG, Garbett KM, White P, Williamson H, Craddock N. Evaluating the effectiveness and acceptability of two positive body image media micro-interventions among children aged 4-6 years old - a study protocol. BMC Public Health. 2024 Dec 19;24(1):3539. doi: 10.1186/s12889-024-20869-z. PMID 39702145